CLINICAL TRIAL: NCT06612918
Title: Effect of High-Intensity Laser Acupuncture on Muscle Performance, Pain, and Quality of Life in Patients With Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of High-intensity Laser Acupuncture on Muscle Performance, Pain and Quality of Life in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005224
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Chronic Nonspecific Low-back Pain
Keywords: low back pain; high-intensity laser acupuncture; muscle performance; back pain; quality of life
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: high-intensity laser acupuncture and exercise therapy program
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity laser acupuncture and the exercise program (Experimental): The patients will receive high-intensity laser acupuncture and the exercise program three times a week for four weeks.
  Interventions: Device: high-intensity laser acupuncture and the exercise program
- sham laser acupuncture and exercises program. (Sham Comparator): The patients will receive sham acupuncture laser and the exercise program three times a week for four weeks.
  Interventions: Other: sham laser acupuncture and the exercises program

INTERVENTIONS:
Device: high-intensity laser acupuncture and the exercise program — The experimental group will receive high-intensity lasers, and the treatment will be performed at 15 acupuncture points: unilateral GV3, GV4, and GV5, and bilateral BL 20, BL23, BL24, BL25, BL40, and GB30. Exercises program: The patients will perform this exercise program in the form of: strengthening exercises for abdominal and back muscles; lumbar stabilization exercises; and stretching exercises.
  Other Names: high-power laser acupuncture
  Arms: high-intensity laser acupuncture and the exercise program
Other: sham laser acupuncture and the exercises program — The patients will receive a sham laser acupuncture and the exercise program in the form of: strengthening exercises for abdominal and back muscles; lumbar stabilization exercises and stretching exercises.
  Other Names: sham laser acupuncture
  Arms: sham laser acupuncture and exercises program.

SUMMARY:
To investigate the effect of high-intensity laser acupuncture on muscle performance, pain, and quality of life in patients with chronic nonspecific low back pain (CNLBP).

DETAILED DESCRIPTION:
Chronic non-specific low back pain (CNSLBP) is a persistent back pain that affects people of all ages and significantly impacts individuals' daily activities and quality of life. While various treatment modalities exist, there is ongoing interest in exploring novel approaches to manage this condition effectively. Laser photobiomodulation (PBM) therapy is a non-invasive and painless method that stimulates cells, pain receptors, and the immune system and can cause analgesic effects. In recent years, high-intensity laser has been used for managing musculoskeletal pain and dysfunction that allows for more energy deposition in deep tissues, resulting in both biological effects and thermal effects. High-intensity laser acupuncture (HILA) has emerged as a promising intervention that combines the therapeutic effects of high-intensity laser therapy and the principles of acupuncture point stimulation on the body (acupoints) to induce physiological effect. However, there is limited evidence supporting HILA efficacy in the management ofCNSLBP, with only a few studies available. For that, this study aims to investigate the effect of HILA on muscle performance, back pain, and quality of life in patients with CNSLBP. Through this current randomized controlled trial, we seek to provide evidence-based insights into the potential effects of this combined approach on measurements of muscle performance, back pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. The patients had CNSLBP with age from 20 to 40 years from both genders.
2. Patients will be referred from an orthopedist with diagnosis of chronic low back pain without underlying pathological causes.
3. The patients with chronic nonspecific low back pain more than 3months. Minimum pain intensity of 30 mm on the visual analogue scale (VAS) for pain, which ranges from 0 to 100 mm.
4. Patients with normal BMI ranges between 18.5:24.9 kg/m2.
5. The study populations must be willing to participate in the study

Exclusion Criteria:

1. Neurological, infectious diseases and systemic illness such as rheumatologic diseases,systemic lupus erythematosus, diabetes mellitus type I or II.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) will also excluded.
4. participation in other treatment within the previous 3 month.
5. Pregnancy.
6. History of spinal fracture, tumor, osteoporosis
7. use of medication, such as corticosteroids, anticonvulsants, and antiinflammatory drugs that may affect the outcome of the study.
8. prior history of adverse effects to physical stimulation therapy.
9. significant physical or mental deficiencies preventing a clear understanding of the study procedure.
10. spinal stenosis, thyroid dysfunctions, obesity, pace-maker.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
muscle performance | up to four weeks]
  Isokinetic dynamometer will be used for measuring muscle performance of back extensors and flexors
muscle performance | follow up after 1 month
  Isokinetic dynamometer will be used for measuring muscle performance of back extensors and flexors

SECONDARY OUTCOMES:
Pain Intensity | up to four weeks
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line.
  Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Pain Intensity | follow up after 1 month
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line.
  Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Quality of Life (WHOQOL-BREF) | up to four weeks
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) will be used in assessment of quality-of-life.The Arabic translation of the WHOQOL-BREF has impressive reliability and validity indices. There will be four domains. The four domain scores will denote an individual perception of quality of life in each particular domain.Domain scores are scaled in a positive direction higher scores denote higher quality of life.
Quality of Life (WHOQOL-BREF) | follow up after 1 month
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) will be used in assessment of quality-of-life.The Arabic translation of the WHOQOL-BREF has impressive reliability and validity indices. There will be four domains. The four domain scores will denote an individual perception of quality of life in each particular domain.Domain scores are scaled in a positive direction higher scores denote higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Giza, Egypt